CLINICAL TRIAL: NCT03862937
Title: Effect of Protein Consumption and Resistance Training on Body Composition, Muscular Strength and Functional Capacity in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Cláudia Dornelles Schneider, Principal Investigator, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FUHSPortoAlegre2019
Record Dates: First submitted 2019-03-03; First posted 2019-03-05 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Elderly; Sarcopenia
Keywords: Protein Supplementation; Body Composition; Resistance Training; Functional Capacity; Muscle Strength
MeSH Terms: conditions — Sarcopenia | interventions — Exercise; Whey Proteins; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The experimental group will perform 12 weeks of strength training twice a week associated with whey protein supplementation.
  Interventions: Dietary Supplement: Exercise training + whey protein
- Placebo (Placebo Comparator): The placebo group will perform 12 weeks of strength training twice a week associated with maltodextrin supplementation.
  Interventions: Other: Exercise training + placebo (maltodextrin)

INTERVENTIONS:
Dietary Supplement: Exercise training + whey protein — Whey protein (2x / day - 20g for breakfast and 20g for dinner).
  Arms: Experimental
Other: Exercise training + placebo (maltodextrin) — Maltodextrin (2x / day - 20g for breakfast and 20g for dinner).
  Arms: Placebo

SUMMARY:
The increase in life expectancy of the world population is associated with a higher incidence of diseases, leading to functional incapacity and dependence in old age. Aging is usually accompanied by progressive loss of muscle mass, muscular strength and functional capacity, possibly exacerbated by inactivity and low protein and energy consumption of elderly individuals. However, the response to strength training, as well as the daily recommendation of protein and other factors related to sarcopenia in this population seem not to be well understood. Objective: To evaluate the effect of protein intake and resistance training on body composition, muscle strength and functional capacity in the elderly. METHODS: A randomized placebo-controlled clinical trial will be conducted with 38 elderly people, ≥ 60 years old, sedentary, and body mass index between 22 and 30 kg / m2. All those who agree to participate will be randomized into two groups (intervention or placebo) and will undergo an initial assessment consisting of food consumption analysis through the application of the three-day food record, assessment of muscle thickness of the thigh and arm by muscle ultrasonography, evaluation of body composition by dual energy X-ray absorptiometry (DEXA), dynamic maximal strength (1RM) test of knee extension and elbow flexion, peak torque test of knee extension, functional capacity tests and quality of life questionnaire (SF-36). The elderly will participate in resistance training for 12 weeks, two session per week. The intervention group will be supplemented with whey protein isolate (2x / day - 20g for breakfast and 20g for dinner) and the placebo group will receive maltodextrin (2x / day - 20g for breakfast and 20g for dinner). All outcomes will be assessed before and after the 12-week resistance training period.

ELIGIBILITY:
Inclusion Criteria:

* Be 60 or older, and in the case of women, they must be postmenopausal (interruption of menstruation for more than one year).
* Have not participated in any systematic exercise program for at least six months prior to the start of this project.
* To have a body mass index (BMI) between 22 and 30 kg / m2.
* Are not cardiopathic, diabetic or have any other metabolic disease.
* Do not present joint problems or any other injury that prevents the proper execution of the exercises of the training routine.
* Non-smoker or have quit smoking for at least five years ago.
* Release of the doctor (medical certificate) to perform the physical exercises.

Exclusion Criteria:

* Do not participate in at least 20 training sessions or miss more than three consecutive training sessions.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-03-03 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Densitometry by dual energy X-ray absorptiometry (DEXA) change from baseline. | This measure will be performed before and after the intervention (12 weeks resistance training and supplementation).
  Measure body composition, such as total fat mass (kg), total fat-free mass (kg), and fat-free mass in the thigh (kg) will be assessed using Dual Energy X-Ray Absorption Densitometry (HXD) (Hologic Discovery W, USA).
Ultrasonography change from baseline. | This measure will be performed before and after the intervention (12 weeks resistance training and supplementation).
  The evaluation of muscle thickness of the quadriceps femoris muscles, as well as the brachial and brachial biceps will be done by means of an image obtained using the Ulio XG ultrasound device (Toshiba, Japan).
Muscular strength (peak of torque) change from baseline. | This measure will be performed before and after the intervention (12 weeks resistance training and supplementation).
  The torque production rate will be calculated from the torque-time curves obtained during a maximal voluntary isometric contraction of knee extension performed on an isokinetic dynamometer (Cybex, Ronkonkoma, USA).
Muscular strength (1-RM) change from baseline. | This measure will be performed before and after the intervention (12 weeks resistance training and supplementation).
  The 1-RM tests (1 maximum repetition test) of knee extension and elbow flexion will be performed in an extensor chair and Scott bench, respectively (Mark Können Gym, China), bilaterally.
Functional capacity (sit and stand up test) change from baseline. | This measure will be performed before and after the intervention (12-week resistance training and supplementation).
  The number of sit and stand movements in the chair will be evaluated in 30 seconds.
Functional capacity (timed up and go test) change from baseline. | This measure will be performed before and after the intervention (12-week resistance training and supplementation).
  The task will be to walk a three-meter course, get around a cone, go back and sit in the chair. The result will be expressed in seconds.
Functional capacity (stair climbing test) change from baseline. | This measure will be performed before and after the intervention (12-week resistance training and supplementation).
  Task to climb a flight of stairs at a comfortable speed and without the aid of the handrail and the time will be measured in seconds.

SECONDARY OUTCOMES:
Protein intake (dietary record) baseline. | To evaluate the food consumption will be used the dietary record of three days.
Protein intake (24-hour food recall). | To verify possible changes in dietary intake over the 12 weeks of intervention, a 24-hour food recall will be applied on the fourth and eighth week and immediately after the last training session.
Diet Quality Index. | To evaluate the quality of the diet will be used the Healthy Eating Index (HEI) that assigns scores to the diet according to the adequacy of the food and nutrients intake, based on the 24 hour reminders previously applied.
Quality of life (SF-36) change from baseline. | This measure will be performed before and after the intervention (12-week resistance training and supplementation). The SF-36 (Medical Outcomes Study 36) questionnaire will be used to evaluate the quality of life of the elderly.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Health Sciences, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No